CLINICAL TRIAL: NCT04638803
Title: A Phase 0, Open-Label, Crossover Microdose Pharmacokinetic Study of PRX-P4-003 In Healthy Volunteers
Brief Title: Microdose Pharmacokinetic Study of PRX-P4-003 In Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Praxis Bioresearch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PBR001; R44116764 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2020-11-04; First posted 2020-11-20 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Prodrugs; Central Nervous System Stimulants

STUDY DESIGN:
Intervention Model Description: In the first arm a fixed order crossover of a PRX-P4-003 followed by administration of the (-)-FCF after a washout period. In the second arm a separate cohort will be administered PRX-P4-003 under fed conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crossover (fasted) (Experimental): On Day 1 subjects are dosed with 100 µg of PRX-P4-003 and PK samples are drawn according to protocol, on Day 15 subjects are dosed with 40 µg of (-)-FCF. Both treatment will be administered under the fasted conditions.
  Interventions: Drug: PRX-P4-003, (-)-FCF
- Single Group (fed) (Experimental): On Day 1 subjects are dosed with 100 µg of PRX-P4-003 and PK samples are drawn according to protocol. The treatment will be administered under the fed condition.
  Interventions: Drug: PRX-P4-003, (-)-FCF

INTERVENTIONS:
Drug: PRX-P4-003, (-)-FCF — sequential study
  Other Names: Prodrug; Stimulant

SUMMARY:
The goal of the present study is to confirm in humans the in-vivo bioconversion of a Prodrug (PRX-P4-003) to (-)-fencamfamine (FCF) the active moiety when orally administered as a single microdose. A second component of the study will evaluate effect of food on pharmacokinetics of PRX-P4-003.

DETAILED DESCRIPTION:
A crossover study comparing blood concentrations after oral administration of microdoses of (-)-fencamfamine (FCF; 40 µg) or its prodrug form (PRX-P4-003; 100 µg)) in the fasted state will be carried out in 4 healthy male volunteers (Study A). This will be followed by determination of blood concentrations of (-)-fencamfamine in a separate cohort of 4 volunteers following oral administration of a microdose of PRX-P4-003 (100 µg) in a fed state (Study B).

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 to 45 years. Willing to fast for at least 8 hours overnight and 4 hours after study drug dose (Study A).
2. BMI within 18 - 32 kg/m2, inclusive.
3. Willing/able to provide signed Informed Consent Form & HIPAA authorization for this study.
4. Agreement to use a highly effective method of birth control with partners of childbearing potential during the study and for 1 month after study dosing such as, abstinence, barrier methods.
5. Normal heart rate (50 to 100 bpm) and blood pressure (diastolic 60-85 mm Hg and systolic 90 to 130 mm Hg, inclusive) at Screening and Day 0.
6. Nonsmoker or has not smoked within the past 6 months of Screening Visit 1 and throughout study participation. Use of recreational and/or medicinal marijuana are NOT permitted within 3 months prior to Screening and during the study. Marijuana use should not be initiated after Screening.
7. Able to communicate well with the Investigator and to comply with the study procedures, requirements, restrictions, and directions of the clinic staff.

Exclusion Criteria:

Main Criteria for Exclusion:

Subjects who meet the following criteria are excluded from study participation

1. History or presence of clinically significant respiratory, GI, renal, hepatic, hematological, neurological (including history of seizure), cardiovascular, psychiatric (including known addictive disorders), musculoskeletal, genitourinary, immunological, or dermatological disorders. The existence of any surgical or medical condition that, in the judgment of the clinical Investigator, might jeopardize the subject's safety, tolerability or interfere with the absorption, distribution, metabolism or excretion of the study drug.
2. Any history of suicide attempts or current suicidal ideation.
3. Abnormal clinically significant laboratory, physical, or neurological findings during screening.
4. Abnormal and clinically significant ECG (as determined by the Investigator or his/her designee) at Screening or Day -0. Abnormalities include, but are not limited to, QTc interval (average of three ECGs) greater than or equal to 450 msec based on 12 lead ECG at Screening or Day -1. Subjects with a history of congenitally prolonged QT interval.
5. In the 14 days (or 5 half-lives, whichever is longer) prior to dosing, the need for prescription medications.
6. Use of acetaminophen greater than a single dose of 1000 mg up to 3 days prior to Day 1.
7. Use of any investigational drug or medical device within 3 months prior to study admission.
8. Known hypersensitivity to, or intolerance of, drugs with the same mechanism of action as PRX-P4-003 or (-)-fencamfamine.
9. Donation or loss of greater than 500 mL of blood in the 8 weeks before dosing. or planned donation of blood at any time during trial participation.
10. History of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) or drug addiction within the past 2 years, as determined by the Investigator. A positive urine drug, or positive alcohol urine (or breath) test at Screening or Day-1.
11. Unwillingness to refrain from alcohol, or illicit or recreational drugs, within 24 hours prior to Day -1and during inpatient period.
12. Seropositive for Hepatitis B, Hepatitis C, (tested during screening) or known HIV infection.
13. The subject is unwilling or unable to comply with the protocol or scheduled appointments.
14. The subject is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male age 18 to 45 years, participants must be willing to fast for 10 hours
Enrollment: 6 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Outcome | 24 hours
  Plasma (-)-FCF exposure (AUC 0-t) after Oral dosing of PRX-P4-003 and (-)-FCF

CONTACTS AND LOCATIONS:
Overall Officials: Kore Liow, MD, Principal Investigator — Hawaii Pacific Neuroscience
Locations (1):
- Hawaii Pacific Neuroscience, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No